CLINICAL TRIAL: NCT03123562
Title: Improvement in Gross Motor Function and Muscle Tone in Children With Cerebral Palsy Related to Neonatal Icterus: An Open-label, Uncontrolled Clinical Trial
Brief Title: Improvement in Gross Motor Function and Muscle Tone in Children With Cerebral Palsy Related to Neonatal Icterus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VinmecRISCGT68
Record Dates: First submitted 2017-04-17; First posted 2017-04-21 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Stem cells; Neonatal icterus
MeSH Terms: conditions — Cerebral Palsy | interventions — Stem Cell Transplantation

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stem cell transplantation (Experimental): Stem cell transplantation 2 intrathecal administrations of autologous bone marrow mononuclear cells at baseline and 6 months afterward
  Interventions: Combination Product: Stem cell transplantation

INTERVENTIONS:
Combination Product: Stem cell transplantation — Transplantation of Autologous Bone Marrow Mononuclear Cells

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of stem cells for cerebral palsy related to neonatal icterus

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and effectiveness of autologous bone marrow mononuclear stem cells in 25 patients with cerebral palsy related to neonatal icterus at Vinmec International Hospital, Hanoi, Vietnam

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy of any types caused by neonatal icterus

Exclusion Criteria:

* Epilepsy
* Hydrocephalus with ventricular drain
* Coagulation disorders
* Allergy to anesthetic agents
* Severe health conditions such as cancer, failure of heart, lung, liver or kidney
* Active infections

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
GMFM-88 and GMFM-66 Percentile | Time Frame: Baseline and 6 months after transplantation
  Change in Total Score of Gross Motor Function Measure GMFM-88 and GMFM-66 Percentile

SECONDARY OUTCOMES:
Change in Muscle tone | Time Frame: Baseline and 6 months after transplantation
  Muscle tone are assessed by Modified Ashworth Scale
Number of adverse events | Through study completion, an average of 6 months
  Examples of adverse events to look for: fever, infections, vomit, epilepsy

CONTACTS AND LOCATIONS:
Overall Officials: Liem T Nguyen, MD., PhD, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nguyen LT, Nguyen AT, Vu CD, Ngo DV, Bui AV. Outcomes of autologous bone marrow mononuclear cells for cerebral palsy: an open label uncontrolled clinical trial. BMC Pediatr. 2017 Apr 12;17(1):104. doi: 10.1186/s12887-017-0859-z. PMID 28403842
- [Result] Jasovic M, Kamenica S, Draganic M, Vasovic P, Nikolajevic A. [Differential diagnosis between mediastinal tumors and aneurysms of the thoracic aorta]. Srp Arh Celok Lek. 1977 Jan;105(1):39-45. No abstract available. Serbian. PMID 905874
- [Derived] Than UTT, Nguyen LT, Nguyen PH, Nguyen XH, Trinh DP, Hoang DH, Nguyen PAT, Dang VD. Inflammatory mediators drive neuroinflammation in autism spectrum disorder and cerebral palsy. Sci Rep. 2023 Dec 18;13(1):22587. doi: 10.1038/s41598-023-49902-8. PMID 38114596
- [Derived] Thanh LN, Trung KN, Duy CV, Van DN, Hoang PN, Phuong ANT, Ngo MD, Thi TN, Viet AB. Improvement in gross motor function and muscle tone in children with cerebral palsy related to neonatal icterus: an open-label, uncontrolled clinical trial. BMC Pediatr. 2019 Aug 22;19(1):290. doi: 10.1186/s12887-019-1669-2. PMID 31438885